CLINICAL TRIAL: NCT07378969
Title: A Non-Interventional Study (NIS) PASS to Characterize Secondary Malignancies of Tcell Origin Following Tisagenlecleucel Therapy (CCTL019B2402)
Brief Title: A Non-Interventional Study PASS to Characterize Secondary Malignancies of Tcell Origin Following Tisagenlecleucel Therapy
Acronym: Lythesia
Status: Not yet recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019B2402
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Secondary Malignancies of T-cell Origin
Keywords: NIS; PASS; secondary malignancies of T-cell origin; tisagenlecleucel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort 1: Individuals who have been treated with tisagenlecleucel in the clinical trial setting but discontinued from the primary interventional study trials, did not move to the long-term follow-up study, or discontinued from the long-term follow-up
- Cohort 2: Cohort 2 includes participants who received tisagenlecleucel in the post-marketing/commercial setting, including patients who received out of specification (OOS) product, or patients enrolled into a MAP (Managed Access Program) or IIT (Investigator Initiated Trial).

SUMMARY:
The study aims to provide an adequate procedural framework to support and facilitate collection of existing participant samples from patients who were diagnosed with secondary malignancy of T-cell origin any time after tisagenlecleucel treatment for testing of muCAR19 transgene and RCL, as well as additional analyses as warranted. Formal testing of existing tumor tissue and/or blood DNA will assess a potential role of tisagenlecleucel in the development/oncogenesis of secondary malignancy of T-cell origin.

DETAILED DESCRIPTION:
The participant population will include individuals who have been treated either in the post-marketing/commercial setting (Cohort 2) or in the clinical trial setting (Cohort 1) but discontinued from the primary interventional study trials, did not move to the LTFU study, or discontinued from the long-term follow-up (LTFU) clinical trial CCTL019A2205B and have a confirmed secondary malignancy of T-cell origin.

The study will remain open for the enrollment of participants from Cohort 1 and Cohort 2 for up to approximately 15 years from the last indication approved for tisagenlecleucel.

ELIGIBILITY:
Inclusion Criteria:

Study participants eligible for inclusion in this study must meet all of the following criteria:

1. Prior use of tisagenlecleucel treatment in CTL019 clinical trial setting or post-marketing/commercial tisagenlecleucel setting as outlined for Cohort 1 and Cohort 2
2. Confirmed diagnosis of secondary malignancy of T-cell origin via redacted pathology report and/or clinical confirmation by the Principal Investigator/clinician responsible for enrolling the participant. Clinical judgement may be required in cases where the diagnosis is not clearly confirmed in the redacted pathology report. There also may be cases in certain site/countries, where sharing the redacted pathology reports is not allowed, hence the clinical diagnosis will be allowed for eligibility.
3. Availability of existing secondary malignancy of T cell origin specimen(s) from tissue, and/or bone marrow aspirate sample(s) and/or blood or DNA extracted from blood (with confirmed T-cell malignancy diagnosis in the sample provided) collected during routine standard of care during the secondary malignancy of T-cell origin diagnosis. Often, only a limited amount of the appropriate sample(s) may be available. For the testing process, a specimen containing the malignant T-cells for the secondary malignancy of T-cell origin must be present. The type of specimen/sample for testing is determined based on the location of the secondary malignancy of T-cell origin. For example, bone marrow aspirate and/or blood and/or bone marrow biopsy may be needed for analysis for a secondary malignancy of T cell origin when the malignant T cells are present in blood and/or bone marrow, and tissue such as a lymph node location or cutaneous or other location is needed when this is the region of the body affected by the secondary malignancy of T-cell origin. Blood, (even if NOT involved with the T cell malignant cells) when available, may also be used for comparison to the tissue/bone marrow used for the analysis. Novartis has established ranges of CAR transgene level in blood for all 3 pivotal trial indications at specific time points. This is used for comparison.

   See laboratory manual for detailed instructions. The following types of samples are recommended for collection if available/pre-existing:
   1. Tumor tissue (FFPE block (ambient temp), unstained slides (ambient temp), or bone marrow aspirate in EDTA or blood in EDTA and frozen, if malignant T-cells present)
   2. Peripheral blood EDTA frozen- to be used when available and either not involved with T-cell malignancy for comparison to the tumor sample provided and/or if peripheral blood has circulating malignant T cells for analysis.
   3. Bone marrow aspirate EDTA frozen if involved with secondary malignancy of T-cell origin.
   4. DNA extracted from blood or bone marrow aspirate stored frozen
   5. Bone marrow biopsy if malignant T-cells are present (FFPE block, unstained slides, ambient temperature)
4. Signed informed consent. For participants who have died, it is acceptable for clinical/academic sites to use a previous biospecimen research consent, or to have an appropriate family member or designated representative to provide consent on behalf of the participant as per local regulations.

Exclusion Criteria:

Study participants meeting any of the following criteria are not eligible for inclusion in this study:

1. Ongoing enrollment on Novartis sponsored CTL019 interventional or LTFU clinical trial
2. Cases where there is no existing available specimens that include the secondary malignancy of T cell origin (tumor tissue and/or existing blood and/or bone marrow and/or DNA from blood for testing)
3. Cases where informed consent is not possible.

Ages: 15 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients who were diagnosed with secondary malignancy of T-cell origin any time after tisagenlecleucel treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2039-08-31 (Estimated); Study Completion 2039-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of muCAR19 qPCR and VCN positive tumors | At screening
  Test specific participant samples using qPCR for muCAR19 transgene/VCN to determine whether the tumor is positive for the muCAR19 transgene with sufficiently positive VCN (≥0.1 viral copies/cell). In cases where there is insufficient DNA to perform qPCR, or when the tumor tissue contains bone (such as bone marrow biopsy), IHC will be performed when feasible. The presence of bone in the sample precludes isolation of DNA of appropriate quality to perform qPCR. In cases where muCAR19 transgene copies are not detectable per qPCR, and/or IHC for muCAR19 is negative, no further testing is performed
Average vector copy number (VCN) and replication competent lentivirus (RCL) among confirmed secondary primary malignancy tumors | At screening
  Average vector copy number (VCN) and replication competent lentivirus (RCL) among confirmed secondary primary malignancy tumors from patients exposed to tisagenlecleucel.
Number of participants with positive muCAR19 IHC and LISA Test | At screening
  For cases where the qPCR for muCART19 is positive in the tumor tissue and the calculated VCN would suggest the presence of a muCAR19 positive tumor, or for positive muCAR19 IHC, LISA will be performed if adequate sample is available

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No